CLINICAL TRIAL: NCT01430650
Title: A Randomised Control Trial to Evaluate Efficacy and Safety of Two Different Protocols of Endometrial Priming for Embryo Transfer.
Brief Title: Endometrial Priming for Embryo Transfer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Miguel Angel Checa, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UREP-PREPENDO-2010
Record Dates: First submitted 2011-06-20; First posted 2011-09-08 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Sterility
Keywords: Oral estrogens; transdermal estrogens; endometrial priming
MeSH Terms: conditions — Infertility | interventions — IDS 89 Sabal serrulata extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral strogen (Experimental)
  Interventions: Drug: Oral strogen
- Transdermal strogen (Experimental)
  Interventions: Drug: Transdermal strogen

INTERVENTIONS:
Drug: Oral strogen — 2 mg of estradiol every day beginning the second day of the cycle until day 7. 4 mg of estradiol every day beginning 8th day of the cycle until day 10. 6 mg of estradiol every day beginning 11th day of the cycle until day 16.
  Arms: Oral strogen
Drug: Transdermal strogen — One patch of 75 mcg of estradiol hemimydrate every 48 h from 2 to day 6. Two patches of 75 mcg of estradiol hemimydrate every 48 h from 6 to day 12. Three patches of 75 mcg of estradiol hemimydrate every 48 h from 12 to day 16.
  Arms: Transdermal strogen

SUMMARY:
The aim of this trial is compare two different endometrial priming protocols

* women that receive oral estrogens
* women that receive transdermal estrogens

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-50 years old with desire of children and needs of embryo transfer.
* Plasma prolactin less than 30.
* Uterine cavity that allow pregnancy, body mass index between 20-30.
* And signed consent inform.

Exclusion Criteria:

* History of estrogen dependent cancer, unknown origin vaginal bleeding.
* Ovarian cyst.
* Contraindications to be pregnant.
* Estrogen allergy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-07; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Difference between day means in endometrial priming to achieve 7 mm. | 11-16 days

SECONDARY OUTCOMES:
Biochemical Pregnancy rate | 26-30 days
  To calculate the biochemical pregnancy rate, we will divide the number of biochemical pregnancy into the number of embryonary transference and multiply by 100.
The patient's adherence to the recommended treatment. | 1-16 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain